CLINICAL TRIAL: NCT01987973
Title: Arthroscopic Repair of Chronic Two-tendon Rotator Cuff Tears by Human Dermal Allograft
Brief Title: Allograft Reconstruction of Massive Rotator Cuff Tears vs Partial Repair Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivan Wong (Other)
Responsible Party: Sponsor-Investigator, Ivan Wong, Orthopedic Surgeon, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-182
Record Dates: First submitted 2013-11-09; First posted 2013-11-20 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Rotator Cuff Syndrome; Rotator Cuff Injury; Disorder of Rotator Cuff; Full Thickness Rotator Cuff Tear; Skin Graft (Allograft) (Autograft) Failure
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Debridement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Partial Repair / Debridement (Active Comparator): Subjects in this arm of the study will receive the intervention "Partial Rotator Cuff Repair". This is the control group.
  Interventions: Procedure: Partial Rotator Cuff Repair
- Allograft Reconstruction (Experimental): Subjects in this arm of the study will receive the intervention "Partial Rotator Cuff Repair with Allograft Augmentation"
  Interventions: Procedure: Partial Rotator Cuff Repair with Allograft Augmentation

INTERVENTIONS:
Procedure: Partial Rotator Cuff Repair — This is the control group. The bursa will be debrided thoroughly and rotator cuff edges will be shaved down to stable tissue. If possible, rip-stop sutures will be employed to stabilize the tear. The subacromial space will then be thoroughly irrigated.
  Other Names: Debridement
  Arms: Partial Repair / Debridement
Procedure: Partial Rotator Cuff Repair with Allograft Augmentation — Patients in this arm will undergo a partial rotator cuff repair (debridement), followed by an allograft augmentation. An Allopatch HD patch will be rehydrated in saline solution for 15 minutes. The patch is then sewn in place with braided polyester suture material. Multiple sutures, approximately 5 to 10 mm apart from one another will be used. The medial sutures are placed at least 3 cm medial to the tendon-bone attachment site. The patch is stretched to remove the manufacturing surface irregularities. The patch is then attached to the greater tuberosity at the tendon-bone attachment site with arthroscopic bone anchors. The subacromial space will then be thoroughly irrigated.
  Other Names: Human dermal allograft; Allograft Reconstruction
  Arms: Allograft Reconstruction

SUMMARY:
The investigators hypothesize that the use of an allograft adjuvant to partial repair will lead to improved shoulder outcome measure scores compared to partial repair alone in massive rotator cuff tears.

DETAILED DESCRIPTION:
A total of 30 patients will be enrolled in the study. Subjects will be randomized into two arms, either (1) Partial Repair/Debridement or (2) Allograft Reconstruction.

The patients will complete a structured clinical examination conducted by a sports medicine fellowship trained orthopaedic consultant, Pre-operatively and Post-operatively at 6 weeks, 3, 6, 12, 24 months. The examination will consist of range of motion testing by goniometer as well as strength testing by hand dynamometer. The patient will also complete the Western Ontario Rotator Cuff Index (WORC) questionnaire.

The main benefit of this procedure is that patients who have currently irreparable massive, chronic rotator cuff tears may acquire a means for their cuff to be repaired. This may aid in improving function of the shoulder, restoring ability to complete activities of daily living, while decreasing pain and sleep disturbances. This would allow the participant to become more functional after rehabilitation. It is our belief that this study could provide new information in helping to understand this relationship, which would in turn lead to future study in this area of orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Large/Massive rotator cuff tear >3cm proven on MRI

Exclusion Criteria:

* Non surgical candidate, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02; Primary Completion 2019-12 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff (WORC) Index | 24 months
  A patient questionnaire evaluating shoulder pain, function.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan H Wong, MD FRCS(C), Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong I, Sparavalo S, King JP, Coady CM. Bridging Allograft Reconstruction Is Superior to Maximal Repair for the Treatment of Chronic, Massive Rotator Cuff Tears: Results of a Prospective, Randomized Controlled Trial. Am J Sports Med. 2021 Oct;49(12):3173-3183. doi: 10.1177/03635465211039846. Epub 2021 Sep 8. PMID 34494901